CLINICAL TRIAL: NCT03072810
Title: Does the Positive Mindfulness Program Increase Wellbeing in People With Chronic Pain?
Brief Title: Positive Mindfulness Program and Wellbeing in Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: University of East London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CanterburyCCU
Record Dates: First submitted 2017-02-20; First posted 2017-03-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Pain, Chronic
Keywords: Positive psychology; Wellbeing; Chronic pain; Mindfulness
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomised wait-list control study
Masking Description: Participants will be aware that they are partaking in the programme and the researcher will see which arm each participant is in. However, participants will be allocated an anonymous code that will be used for storing and analysing outcome data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive mindfulness program (Experimental): Participants will receive a 4 week online positive mindfulness program as described in previous sections.
  Interventions: Behavioral: Positive mindfulness program
- Waitlist control (Other): Participants will receive the same intervention as the intervention arm (positive mindfulness program) but will be required to wait 4 weeks before commencing.
  Interventions: Behavioral: Positive mindfulness program

INTERVENTIONS:
Behavioral: Positive mindfulness program — 4 week program consisting of 8 modules. Each module comprises an introduction video (approx. 10 minutes), a daily meditation (approx. 10 minutes) and a daily activity.

SUMMARY:
This study aims to increase the well-being of individuals with chronic pain through a 4-week online positive mindfulness programme. Each module, lasting 4 days, will include a daily meditation and focus on a different aspect of positive psychology. This is a quantitative study. The independent variable is participation in the programme. The dependent variables are: wellbeing, mindfulness, pain severity, pain catastrophising and health quality of life. There will be one experimental group who participate in the programme as soon as they are recruited. There will be one control group who are put on a 'wait-list' to complete the programme after an 8 week wait. Pre and post measures will be taken. Participants are being recruited through NHS clinics in London and Oxford, including the Pain Management Centre at Oxford University Hospitals (Churchill site) and INPUT at St Thomas's Hospital (which are participant identification centres). Participants who hear about the study via other means including online or through word of mouth are also being accepted.

DETAILED DESCRIPTION:
Practicing mindfulness has been demonstrated to have a variety of benefits such as reducing stress, depression, anxiety, insomnia and pain symptoms. Positive psychology interventions have been shown to increase well-being by enhancing resilience, improving health and having a positive impact on levels of anxiety and depression.

The clinical guidance for treating individuals with chronic pain recommends reducing stress and improving sleep and supporting patients to gain a greater sense of control over their illness. Mindfulness has been shown to be effective in supporting patients with chronic pain to achieve these outcomes.

This study is the first of its kind to combine aspects of positive psychology and mindfulness to create an online programme specifically designed to enhance well-being. Previous participants who have undertaken the Positive Mindfulness Programme have experienced reduced depression and stress and an increase in well-being.

Participants will be recruited through the Pain Management Centre at Oxford University Hospitals (Churchill site) and INPUT at St Thomas's Hospital. Patients with chronic pain will be asked by their clinician if they would like to participate in the study. Clinicians will then pass on (with consent) the contact details of interested potential participants to the researcher. Patients can alternatively choose to get in touch with the researcher directly themselves. Participants will undertake the online programme independently in any location they choose to access the programme.

All participants will be sent an introductory email with a link to an online survey platform where they will be asked to complete 5 pre-validated questionnaires. Within this invitation email, the structure of the programme and daily commitment will be described. The researcher's contact details will be provided should potential participants have any questions regarding the 4-week programme. Participants will be asked to sign an online consent form as part of the initial completion of the outcome measures, before they commence the programme. Participants will logon to the online platform by creating a personalised, anonymous username and password.

Once the participants have completed the baseline outcome measures, the experimental group will be sent a link to the Positive Mindfulness Programme online course and they will be able to begin the 4 week course. Participants will have controlled access to the website so will be unable to start earlier than their slot.

Each week participants will watch a short video providing the theoretical basis for the aspect of Positive Psychology and mindfulness they will be practicing. Each video will be between 8 - 10 minutes long. At the end of the theory video, participants are asked to access and download an audio file which provides them with their daily meditation practice for the week. The audio files containing the daily meditation lasts 12-15 minutes. At the end of each meditation, participants are invited to engage in a daily activity that has a positive psychology focus. The topics covered include: self-awareness, positive emotions, self-compassion, autonomy, self-efficacy, meaning, relations with others and engagement.

Participants are asked to practice the meditation daily. After practicing the meditation for 4 days, participants will log back into the survey site to complete the next week's material. Participants continue this same process for the duration of the 4-weeks.

Upon completion of the 4 weeks of material, participants will be given a wrap-up session that summarises each week of the programme. They will then be asked to complete the same questionnaires that were administered at the beginning of the programme, thus providing post-measures. One month after completion, participants will be contacted again to complete the same series of questions.

Throughout the programme there will be a control group. This group will be asked to complete the same measures at the same time points as the study group (immediately, at 4 weeks, at 8 weeks). However, these individuals will not participate in the weekly programme until 8 weeks has passed. Once they have waited 8 weeks they will be offered the 4 week programme.

ELIGIBILITY:
Inclusion Criteria:

* Is experiencing chronic pain that has lasted for at least 3 months at time of entry to study
* Has access to the internet daily

Exclusion Criteria:

* Currently receiving another form of psychological intervention
* Post Traumatic Stress Disorder
* Eating disorders
* Substance abuse (inc prescription drugs)
* Subjected to torture or abuse Suspected factitious illness or dissociative symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change in mindfulness (using Freiburg Mindfulness Inventory) | Baseline, 4 weeks, 8 weeks
  This 14 item scale measures mindfulness and will be used to check whether the intervention increases mindfulness.
Change in wellbeing (using PERMA profiler) | Baseline, 4 weeks, 8 weeks
  Developed by Butler and Kern (2015). The scale measures the five aspects of the PERMA theory of wellbeing (Seligman, 2011).

SECONDARY OUTCOMES:
Change in pain catastrophizing (using Pain Catastrophizing Scale) | Baseline, 4 weeks, 8 weeks
  (Sullivan, Bishop and Pivik, 1995). A 13 item scale that measures overall level of catastrophizing about pain and provides sub-scores on the components of rumination, magnification and helplessness.
Change in subjective pain levels (using Symptom severity and widespread pain index) | Baseline, 4 weeks, 8 weeks
  (Hauser et al., 2012). The measure has high correlation with the PHQ-4 and good criterion validity when compared against the Fibromyalgia diagnostic criteria.
Change in health quality of life (using EQ-5D-5L) | Baseline, 4 weeks, 8 weeks
  (Health Quality of Life Questionnaire; Herdman et al., 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lavender, Professor, Study Director — Canterbury Christ Church University; Itai Ivtzan, Dr, Principal Investigator — University of East London; Abi Davison Jenkins, DClinPsy, Principal Investigator — Canterbury Christ Church University
Locations (3):
- United Kingdom (3):
  - Canterbury Christ Church University, Royal Tunbridge Wells, Kent
  - Churchill Hospital, Oxford, Oxfordshire
  - INPUT, St Thomas's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walach, H., Buchheld, N., Buttenmüller, V., Kleinknecht, N., & Schmidt, S. (2006). Measuring mindfulness-the Freiburg mindfulness inventory (FMI). Personality and Individual Differences, 40(8), 1543-1555.
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Hauser W, Jung E, Erbsloh-Moller B, Gesmann M, Kuhn-Becker H, Petermann F, Langhorst J, Weiss T, Winkelmann A, Wolfe F. Validation of the Fibromyalgia Survey Questionnaire within a cross-sectional survey. PLoS One. 2012;7(5):e37504. doi: 10.1371/journal.pone.0037504. Epub 2012 May 25. PMID 22662163
- [Background] Butler, J. and Kern, M. (2015, September 25). The PERMA Profiler. Retrieved from http://www.peggykern.org/uploads/5/6/6/7/56678211/the_perma-profiler_092515.pdf
- [Background] Sullivan, M. J., Bishop, S. R., & Pivik, J. (1995). The pain catastrophizing scale: development and validation. Psychological assessment, 7(4), 524.
- [Background] Ivtzan, I. (2015). Positive Mindfulness Program (Chronic Pain). Retrieved from http://www.awarenessisfreedom.com/courses/positive-mindfulness-program-chronic-pain/
- [Background] Ivtzan, I. (2015). Integrating Mindfulness in Positive Psychology: A Randomised Controlled Trial of an 8-week Positive Mindfulness Programme (PMP). Manuscript submitted for publication.